CLINICAL TRIAL: NCT05579639
Title: Reduction of Bloodstream Infections From Oral Organisms in Pediatric Stem Cell Transplant: a Randomized, Multicenter, Double-blind , Placebo-controlled Study Evaluating Twice Daily Oral Xylitol
Brief Title: Xylitol BSI Multisite - Reduction of Bloodstream Infections From Oral Organisms in Pediatric Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-0537; 1UG3DE030401-01 (NIH)
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Allogeneic Stem Cell Transplantation
Keywords: bloodstream infections; oral health; xylitol; dental health; gingivitis; mucositis; plaque
MeSH Terms: conditions — Sepsis; Gingivitis; Mucositis; Plaque, Amyloid | interventions — Xylitol

STUDY DESIGN:
Intervention Model Description: randomized, multicenter, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, parents/guardians, nursing staff (interventionists), oral evaluators, and investigators will be blinded to the intervention, administered in the form of twice-daily grape-flavored xylitol wipes or grape-flavored saline wipes (controls). Preformed packets will be prepared by CCHMC Investigational Pharmacy staff, which will consist of either saline wipes with natural grape flavoring or xylitol. The color, taste, and smell of the wipes will be identical. The statistician will be unblinded to treatment assignment for the analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xylitol (Experimental): Xylitol, a naturally occurring sugar alcohol found in plums, strawberries, and various vegetables such as cauliflower, has been approved for use in food by the US FDA since 1963. Spiffies Xylitol Wipes will be used.
  Interventions: Other: Xylitol
- Grape-flavored Wipes (Placebo Comparator): Grape-flavored wipes will be used with 2 drops of PCCA colorless grape flavoring. The grape-flavored wipes each contain a solution of 0.9% Sodium Chloride, purified water, and Benzalkonium chloride. PCCA artificial colorless grape flavoring will be used. The PCCA grape flavoring contains propylene glycol, ethyl alcohol, and artificial flavoring.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Xylitol — Xylitol wipes
  Other Names: Spiffies Xylitol Wipes
  Arms: Xylitol
Other: Placebo — Placebo wipes
  Other Names: Grape-Flavored Wipes
  Arms: Grape-flavored Wipes

SUMMARY:
Bloodstream infections (BSI) caused by bacteria translocating across injured oral mucosa are a significant cause of morbidity and mortality in patients undergoing stem cell transplantation (SCT). Unfortunately, there are currently no known strategies to prevent these BSI in this vulnerable population. The investigators will conduct a randomized, double-blind, placebo-controlled trial at three institutions to evaluate the effectiveness of twice daily intraoral xylitol-wipe application on reducing BSI in pediatric SCT patients.

DETAILED DESCRIPTION:
Patients will be randomized to receive either twice-daily intraoral grape-flavored xylitol-wipe (intervention arm) or grape-flavored saline wipe (control arm) application in addition to the current standard of care (SOC). The purpose of this study is to determine whether xylitol wipes are effective at reducing bloodstream infections (BSIs), dental plaque, mucositis (redness and ulcers in the mouth), or gingivitis in patients who undergo allogeneic stem cell transplant (SCT).

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent and assent (when applicable) form
* Willing to comply with all study procedures and be available for the duration of the study
* Admitted and planning to undergo an allogeneic stem cell transplant (SCT) at Cincinnati Children's Hospital Medical Center (CCHMC), Boston Children's Hospital, or Children's Hospital of Colorado (Denver).
* Male or female, 4 months to 25 years of age at the time of SCT (Day 0)
* Have a minimum of one tooth
* Agree to avoid chewing gum and toothpaste that contains xylitol during the intervention period

Exclusion Criteria:

* Prior radiation treatment for cancer of the oral cavity, head, or neck in the past 6 months per the study participant's medical record
* Cranial boost in patients receiving total body irradiation
* Known history of allergy to xylitol
* Known history of allergy to grapes or grape flavoring
* Undergoing a conditioning-free allogeneic stem cell transplant (patient does not receive any chemotherapy or radiation prior to stem cell infusion)

Ages: 4 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 419 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Bacteremia from an oral organism | 33 days
  Incidence of bloodstream infection (BSI) from oral flora organisms in in patients receiving xylitol compared to placebo

SECONDARY OUTCOMES:
Bacteremia from other non-oral flora organisms | 33 days
  Incidence of BSI from non-oral flora organisms in patients receiving xylitol compared to placebo
Dental plaque | 33 days
  Debris Index Simplified (DI-S) score
Gingivitis | 33 days
  Mean Modified Gingival Index (MGI) score
Objective mucositis | 33 days
  Mean Oral Mucositis Assessment Scale (OMAS) score
Patient-reported mucositis | 33 days
  ChIMES total score
Oral microbiome diversity | 33 days
  Shannon Diversity Index

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dandoy, MD, MSc, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Dana-Farber/Boston Children's, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No